CLINICAL TRIAL: NCT02445534
Title: Registry of Cell Therapy in Non-Ischemic Dilated Cardiomyopathy
Acronym: RECORD
Status: Recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Bojan Vrtovec, Medical Director, Advanced Heart Failure and Transplantation Center, University Medical Centre Ljubljana
Other Study IDs: RECORD
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Cardiomyopathy, Dilated
Keywords: Cell Therapy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Autologous stem cell therapy — All patients received granulocyte-colony stimulating factor (G-CSF; 5 mg/kg, 5 days). CD34+ cell were then collected by apheresis and injected transendocardially or intracororonary.

SUMMARY:
Although several studies have demonstrated beneficial effects of stem cell therapy in patients with non-ischemic dilated cardiomyopathy, the long term benefits and predictors of response to therapy remain undefined. The aim of this registry is to pool long-term clinical data in patients with non-ischemic dilated cardiomyopathy undergoing autologous cell therapy in an attempt to better define predictors of response to such treatment.

DETAILED DESCRIPTION:
Registry will include all patients who underwent intracoronary or intramyocardial cell therapy as a part of clinical trials performed at UMC Ljubljana from January 2005 until January 2018. Patients will be followed on regular basis in a dedicated heart failure outpatient clinic, clinical data will be collected and stored in a secure central database. Data will be analyzed in periodic intervals by an independent Data monitoring board in an attempt to better define the predictors of clinical response to cell therapy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria consisted of the following: age 18-65 years old, diagnosis of DCM according to the European Society of Cardiology position statement (9), optimal medical management for at least 6 months, left ventricular ejection fraction (LVEF) <40%, and New York Heart Association functional Class III on stable medical therapy for at least 3 months before referral.

Exclusion Criteria:

* Patients with acute multi-organ failure or a history of hematologic neoplasms were not included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled in clinical trials of stem cell therapy in non-ischemic dilated cardiomyopathy at UMC Ljubljana from January, 2005 will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2005-01; Primary Completion 2027-01 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Transplantation-free survival | 5 years
  Survival after 5 years without undergoing heart transplantation

SECONDARY OUTCOMES:
Changes in left ventricular ejection fraction | 5 years
Changes in left ventricular dimensions | 5 years
Changes in left ventricular diastolic function | 5 years
Changes in right ventricular function | 5 years

OTHER OUTCOMES:
Changes in exercise capacity | 5 years
Changes in NT-proBNP | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Vrtovec, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Frljak S, Poglajen G, Zemljic G, Cerar A, Haddad F, Terzic A, Vrtovec B. Larger End-Diastolic Volume Associates With Response to Cell Therapy in Patients With Nonischemic Dilated Cardiomyopathy. Mayo Clin Proc. 2020 Oct;95(10):2125-2133. doi: 10.1016/j.mayocp.2020.02.031. PMID 33012343
- [Derived] Bervar M, Kozelj M, Poglajen G, Sever M, Zemljic G, Frljak S, Cukjati M, Cernelc P, Haddad F, Vrtovec B. Effects of Transendocardial CD34+ Cell Transplantation on Diastolic Parameters in Patients with Nonischemic Dilated Cardiomyopathy. Stem Cells Transl Med. 2017 Jun;6(6):1515-1521. doi: 10.1002/sctm.16-0331. Epub 2017 Mar 11. PMID 28296283